CLINICAL TRIAL: NCT05711160
Title: Accuracy and Reliability of Teeth Widths and Bolton' Ratios Measured in Cone-Beam Computer Tomography and Intra Oral Scanner Images Compared With Plaster Models (Gold Standard) in a Sample of Duhok Population.
Brief Title: Comparison of the Accuracy and Reliability of Measurements Made on CBCT and IOS Images With Their made-on Plaster Models.
Status: Completed | Type: Observational
Sponsor: University of Duhok (Other)
Responsible Party: Principal Investigator, Mohamad Radwan Sirri, Study Director-Iraq-Duhok, University of Duhok
Other Study IDs: SL1990
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Malocclusion
Keywords: plaster model; cone beam computed tomography.; intraoral scanner; teeth widths; Bolton' ratios.; CBCT; IOS
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malocclusion patients: Patients with different types of malocclusion will be included. Plaster models will be fabricated after pouring the impressions with hard gypsum.
  All patients have been undergoing CBCT scans for both jaws. Then, intraoral scanned of the dental arches of each patient have been taken using an intraoral scanner. Then measurements were made on digital images (CBCT & IOS) and on plaster models.
  Interventions: Diagnostic Test: Plaster models; Diagnostic Test: CBCT images; Diagnostic Test: IOS images

INTERVENTIONS:
Diagnostic Test: Plaster models — The impressions taken of the dental arches will be poured with hard gypsum in order to make use of the models for taking measurements. These measurements will be considered the gold standard.
  Other Names: Study models; Study casts; Poured study models
Diagnostic Test: CBCT images — All patients have been undergoing CBCT scans for both jaws
  Other Names: cone beam computed tomography images.
Diagnostic Test: IOS images — The patient's teeth have been dried with air syringe and scanned with the Intraoral scanner
  Other Names: intra oral scanner images

SUMMARY:
The orthodontist uses plaster models to collect information. This includes identification deviations, classification of malocclusion, formulation of treatment goals for specific patient. Models are used to examine the morphology of individual teeth and also to visualize the placement of teeth in individual dental arches. Study models It therefore appears to be one of the most important records for treatment planning.

In USA, orthodontist can start practicing orthodontics which requires a lot of difficulty 300 new cases in a year and therefore may require an entire room to store plaster models. The minimum file retention period depends on the appropriate platform for the statute of limitations during which legal action for fault can be brought. in the USA, this time period varies from 5 to 15 years, varies from country to country.

This platform can be started on the last day of treatment, or it can be postponed until the patient reaches adulthood. Regardless of how it is viewed, long term storage is required. Over ten years, if 300 new cases are initiated each year, that will represent 6,000 combinations of prototyping, pre-processing and post-processing. Additional storage space may be required, maybe somewhere else, with financial implications.

With the recent introduction of digital models and CBCT images, the orthodontist now has an alternative to traditional plaster study models. Digital technology makes it possible to analyze a computer using software capable of rotating, examining and measuring digital images of the model and dental arches from different points of view. The intraoral scanner is a hand-held device that creates digital impressions of the oral fossa and displays it in 3D on a computer screen after being processed by the scanning program for each device. By 1985 the first intraoral scanner was available for commercial use, and over time it had evolved to become smaller, faster, and more accurate. Intraoral scanners provide easier treatment planning, better workflow, greater patient acceptance and shorter working time, but more studies are needed to investigate their accuracy and compare with traditional methods. The measurements of the tooth widths are one of the important elements in orthodontic diagnosis because of its role in calculating the partial and total Bolton ratio, the Ton relationship, and space analysis. Therefore, the aim of this study will be to assess the accuracy and reliability of measuring teeth widths and Bolton ratios based on three mains well -known methods (plaster models, CBCT images and intraoral images) to ensure the safety of orthodontic diagnostic outputs.

DETAILED DESCRIPTION:
Several published studies analyzed teeth widths and Bolton' ratios using CBCT with plaster models, two-dimensional images, or three-dimensional images as the gold standard and applied to patients or skulls, but they did not use the sagittal axis orientation method for each tooth on the limit to determine its precise lateral mesial width, but the method of unified orientation was adopted in the transverse plane.

The most important benefit of the CBCT is that the measurements are made directly on the digital model, which eliminates the possibility of error that can occur with traditional methods (alginate blending, alginate hardening, casting) or some other digital methods (such as scanning plaster model).

The special orientation method was adopted for each tooth separately so that the three axes of the software are perpendicular to the longitudinal axis of the tooth, and the maximum mesio-lateral width is determined on both the axial plane and the transverse plane, and the measurement is made on each of them, which is supposed to be identical in the case of correct orientation.

This method is useful for determining the width of each tooth, regardless of its position within the dental arch or overlapping it with other teeth.

The intraoral scan is the latest innovation in dentistry to generate three-dimensional models that can be studied, and many tests were conducted on it to determine its accuracy and reliability by determining teeth widths and the Bolton ratios with the adoption of plaster models or two-dimensional images as a gold standard.

Looking at the published medical literature, and in an attempt to find a study similar to the current study, It was found that the comparisons regarding teeth widths measurements were among plaster models (as a gold standard) and CBCT images or between plaster models (as a gold standard) and IOS images, and no study was found that made a comparison Triple among the previous three methods.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 35 years.
2. Full permanent dentition from right first molar to left first molar in both upper and lower arches.
3. Participants should not be under orthodontic treatment.

Exclusion Criteria:

1. Tooth agenesis or extractions.
2. Presence of large restorations that could change the mesiodistal diameters of the teeth.
3. Teeth with anomalous shapes.
4. Teeth with large carious lesions.
5. Enamel defects that affect the morphology of crown.
6. Severe crowding in the dentition (< 6 mm).
7. Missing or heavily restored teeth.
8. Teeth with large carious lesions / enamel defects that affect the morphology of crown/

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with different levels of malocclusion
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Tooth width using plaster models. | After seven days of taking the impressions of the dental arches. Silicon Impressions have been taken in the same day of patient's entry to the study
  Maximum mesiodistal width of each crown (from the first molar to the first molar of each jaw) has been measured between the anatomic contact areas when the teeth will correctly align using a digital electronic caliper. The result is expressed in mm.
Tooth width using CBCT images. | After seven days of taking the CBCT scans for both jaws. CBCT images have been taken in the same day of patient's entry to the study.
  For the anterior teeth: (centrals, laterals and canines) On the cross section & frontal section: Maximum mesiodistal width of each crown (from the first molar to the first molar of each jaw) has been measured between the anatomic contact point.
  The result is expressed in mm. For the posterior teeth: (premolars and first molars) On the cross section & sagittal section: Maximum mesiodistal width of each crown (from the first molar to the first molar of each jaw) has been measured between the anatomic contact point.
  The result is expressed in mm. This method was adopted to obtain the true width of each tooth, regardless of its position within the dental arch.
Tooth width using IOS images. | After seven days of scanned with the Intraoral scanner for both jaws. IOS images have been taken in the same day of patient's entry to the study
  Digital images have been opened in the software, and Maximum mesiodistal width of each crown (from the first molar to the first molar of each jaw) has been measured between the anatomic contact point using the "Diagnostics" tool.
Anterior Bolton' ratio using plaster models. | After seven days of taking the impressions of the dental arches. Silicon Impressions have been taken in the same day of patient's entry to the study
  Bolton analysis is used to identify disharmony between maxillary and mandibular tooth size which is considered an important factor to ensure the success of orthodontic treatment. With the application of the suggested formula, the partial ratio should be 77.2% (±1.65) The formula is the sum of the mesio-distal widths of the lower six anterior teeth divided by the sum of the mesio-distal widths of the upper six anterior teeth.
Anterior Bolton' ratio using CBCT images. | After seven days of taking the CBCT scans for both jaws. CBCT images have been taken in the same day of patient's entry to the study.
  Bolton analysis is used to identify disharmony between maxillary and mandibular tooth size which is considered an important factor to ensure the success of orthodontic treatment. With the application of the suggested formula, the partial ratio should be 77.2% (±1.65) The formula is the sum of the mesio-distal widths of the lower six anterior teeth divided by the sum of the mesio-distal widths of the upper six anterior teeth.
Anterior Bolton' ratio using IOS images. | After seven days of scanned with the Intraoral scanner for both jaws. IOS images have been taken in the same day of patient's entry to the study
  Bolton analysis is used to identify disharmony between maxillary and mandibular tooth size which is considered an important factor to ensure the success of orthodontic treatment. With the application of the suggested formula, the partial ratio should be 77.2% (±1.65) The formula is the sum of the mesio-distal widths of the lower six anterior teeth divided by the sum of the mesio-distal widths of the upper six anterior teeth.
Overall Bolton' ratio using plaster models. | After seven days of taking the impressions of the dental arches. Silicon Impressions have been taken in the same day of patient's entry to the study
  Bolton analysis is used to identify disharmony between maxillary and mandibular tooth size which is considered an important factor to ensure the success of orthodontic treatment. With the application of the suggested formula, the overall ratio should be 91.3%. The formula is the sum of the mesio-distal widths of the lower twelve teeth divided by the sum of the mesio-distal widths of the upper twelve teeth.
Overall Bolton' ratio using CBCT images. | After seven days of taking the CBCT scans for both jaws. CBCT images have been taken in the same day of patient's entry to the study.
  Bolton analysis is used to identify disharmony between maxillary and mandibular tooth size which is considered an important factor to ensure the success of orthodontic treatment. With the application of the suggested formula, the overall ratio should be 91.3%. The formula is the sum of the mesio-distal widths of the lower twelve teeth divided by the sum of the mesio-distal widths of the upper twelve teeth.
Overall Bolton' ratio using IOS images. | After seven days of scanned with the Intraoral scanner for both jaws. IOS images have been taken in the same day of patient's entry to the study
  Bolton analysis is used to identify disharmony between maxillary and mandibular tooth size which is considered an important factor to ensure the success of orthodontic treatment. With the application of the suggested formula, the overall ratio should be 91.3%. The formula is the sum of the mesio-distal widths of the lower twelve teeth divided by the sum of the mesio-distal widths of the upper twelve teeth.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamad Radwan Sirri, Duhok, Iraq

REFERENCES:
- [Result] Kim J, Lagravere MO. Accuracy of Bolton analysis measured in laser scanned digital models compared with plaster models (gold standard) and cone-beam computer tomography images. Korean J Orthod. 2016 Jan;46(1):13-9. doi: 10.4041/kjod.2016.46.1.13. Epub 2016 Jan 25. PMID 26877978
- [Result] Paredes V, Gandia JL, Cibrian R. Determination of Bolton tooth-size ratios by digitization, and comparison with the traditional method. Eur J Orthod. 2006 Apr;28(2):120-5. doi: 10.1093/ejo/cji077. Epub 2005 Dec 22. PMID 16373454
- [Result] Wiranto MG, Engelbrecht WP, Tutein Nolthenius HE, van der Meer WJ, Ren Y. Validity, reliability, and reproducibility of linear measurements on digital models obtained from intraoral and cone-beam computed tomography scans of alginate impressions. Am J Orthod Dentofacial Orthop. 2013 Jan;143(1):140-7. doi: 10.1016/j.ajodo.2012.06.018. PMID 23273370
- [Result] Kumar AA, Phillip A, Kumar S, Rawat A, Priya S, Kumaran V. Digital model as an alternative to plaster model in assessment of space analysis. J Pharm Bioallied Sci. 2015 Aug;7(Suppl 2):S465-9. doi: 10.4103/0975-7406.163506. PMID 26538899
- [Result] Alam MK, Shahid F, Purmal K, Ahmad B, Khamis MF. Bolton tooth size ratio and its relation with arch widths, arch length and arch perimeter: a cone beam computed tomography (CBCT) study. Acta Odontol Scand. 2014 Nov;72(8):1047-53. doi: 10.3109/00016357.2014.946967. Epub 2014 Sep 15. PMID 25220521